CLINICAL TRIAL: NCT04516369
Title: An Open-label, Single-arm Study to Provide Efficacy and Safety Data of Voretigene Neparvovec Administered as Subretinal Injection in Japanese Patients With Biallelic RPE65 Mutation-associated Retinal Dystrophy
Brief Title: Study of Efficacy and Safety of Voretigene Neparvovec in Japanese Patients With Biallelic RPE65 Mutation-associated Retinal Dystrophy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTW888A11301; 2019-003781-41 (EudraCT Number)
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Biallelic RPE65 Mutation-associated Retinal Dystrophy
Keywords: LTW888; voretigene neparvovec; Biallelic RPE65 mutation-associated retinal dystrophy; Japanese patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voretigene neparvovec (Experimental): 1.5 E11 vg (0.3 mL subretinal injection in each eye, 6-18 days apart)
  Interventions: Genetic: voretigene neparvovec

INTERVENTIONS:
Genetic: voretigene neparvovec — Voretigene neparvovec is an adeno-associated viral type 2 (AAV2) gene therapy vector driving expression of normal human retinal pigment epithelium 65 kDa protein (hRPE65) gene.

SUMMARY:
The purpose of this study is to provide safety and efficacy data for voretigene neparvovec, administered as subretinal injection, in Japanese patients with biallelic RPE65 mutation-associated retinal dystrophy.

DETAILED DESCRIPTION:
This is an open-label, single-arm study to evaluate the safety and efficacy of bilateral subretinal administration of voretigene neparvovec in Japanese patients with biallelic RPE65 mutation-associated retinal dystrophy. Assessments will include full-field light sensitivity threshold testing, visual fields, visual acuity, vector shedding, immunogenicity and adverse events. Participants will be monitored for 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants with biallelic RPE65 mutation-associated retinal dystrophy; molecular diagnosis of RPE65 mutation must be confirmed by a Novartis designated laboratory in Japan.
* Age four years or older.
* Visual acuity worse than 20/60 (both eyes) and/or visual field less than 20 degrees in any meridian as measured by a III4e isopter or equivalent (both eyes).
* Sufficient viable retinal cells as determined by non-invasive means, such as optical coherence tomography (OCT) and/ or ophthalmoscopy. Must have either:

  * An area of retina within the posterior pole of > 100 µm thickness shown on OCT, or
  * ≥ 3 disc areas of retina without atrophy or pigmentary degeneration within the posterior pole, or
  * Remaining visual field within 30 degrees of fixation as measured by a III4e isopter or equivalent

Exclusion Criteria:

* Any prior participation in a study in which a gene therapy vector was administered.
* Participation in a clinical study with an investigational drug in the past 6 months from screening visit.
* Known hypersensitivity to any of the study treatments including excipients or to medications planned for use in the peri-operative period.
* Unable to reliably perform the FST assessment.
* Use of retinoid compounds or precursors that could potentially interact with the biochemical activity of the RPE65 enzyme in the past 6 months from screening visit.
* Prior intraocular surgery within 6 months from screening visit.
* Prior use of any medicines that, in the opinion of the investigator, may have caused retinal damage (e.g., sildenafil or related compounds, hydroxychloroquine, chloroquine, thioridazine, any other retino-toxic compounds)
* Pre-existing eye conditions or complicating systemic diseases that would preclude the planned surgery or interfere with the interpretation of study. Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter ocular function.

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in full-field light sensitivity threshold | Baseline, Day 30, 90, 180, 270, and Year 1 after second eye injection
  Full-field light sensitivity threshold (FST) is evaluated using white light, as averaged over both eyes.

SECONDARY OUTCOMES:
Change from Baseline in visual field | Baseline, Day 14, 30, 90, 180, 270, and Year 1, 2, 3, 4, 5 after second eye injection
  Visual Field is assessed using the sum total degrees for VF, averaged over both eyes, as measued using Goldmann kinetic perimetry testing with a III4e target.
Change from Baseline in macular threshold | Baseline, Day 14, 30, 90, 180, 270, and Year 1, 2, 3, 4, 5 after second eye injection
  Macular threshold is assessed as averaged over both eyes, as measured using Humphrey static visual field testing.
Change from Baseline in visual acuity | Baseline, Day 1, and 3 after first eye injection; Day 1, 3, 14, 30, 90, 180, 270, and Year 1, 2, 3, 4, 5 after second eye injection
  Visual acuity is assessed as averaged over both eyes.
Change from Baseline in FST for long-term period | Baseline, Year 2, 3, 4 and 5 after second eye injection
  FST is assessed using white light, as averaged over both eyes.
Proportion of subject with the presence of vector shedding of voretigene neparvovec during the study period | Baseline, Day 0, 1 and 3 after first eye injection; Day 0, 1, 3, 14, 30, 90, 180, 270, and Year 1 after second eye injection
  Assessed as the presence of vector in peripheral blood or collected tear.
Proportion of subject with the presence of immunogenicity of voretigene neparvovec during the study period | Baseline, Day 30, 90, 180, 270, and Year 1 after second eye injection
  Assessed as presence of systemic cell-mediated or humoral responses to capsid or transgene product .

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Meguro-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com